CLINICAL TRIAL: NCT05360472
Title: Evaluation of Feconomics Versus Traditional Techniques for Diagnosis of Intestinal Parasitic Infections
Brief Title: Evaluation of Feconomics for Diagnosis of Intestinal Parasitic Infections
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shorouk Nasser Mahmoud, Demonstrator at medical parasitology department, Faculty of medicine, Sohag University
Other Study IDs: soh-med-22-04-17
Record Dates: First submitted 2022-04-28; First posted 2022-05-04 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Intestinal Parasitic Infection
MeSH Terms: conditions — Intestinal Diseases, Parasitic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stool specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People of all ages are affected by intestinal parasitic infections(IPIs) ; however, children are the most commonly affected, which is linked to their poor hygienic practices, and weak immune status. In children, IPIs are associated with malabsorption, weight loss, anemia, poor growth rate, learning difficulties, mental retardation and intellectual problems . The difficulty of diagnosis is the main problem in the control of intestinal parasitic infections. The choice of a particular technique is usually influenced by affordability, simplicity, cost, sensitivity in addition to the level of technical skills involved. Microscopic examination remains the cornerstone of parasitological diagnosis which is time consuming and requires an experienced observer to identify the organism. Formalin-ether sedimentation technique is commonly used in laboratories owing to its ability to isolate a large variety of parasites. However, it's a labor intensive procedure and is usually associated with hazards of using the inflammable lipid solvents. The drawbacks of the previous techniques have encouraged the development of commercial products such as Feconomics which is a new ready to use kit for concentration of stool samples in parasitological diagnosis.

The aim of the study is :

evaluation of the efficacy of Feconomics technique in comparison to traditional techniques i.e., direct smear and formalin ethyl acetate sedimentation technique for the diagnosis of intestinal parasites in school children.

ELIGIBILITY:
Inclusion Criteria:

* school children whose age is between 6-12 years

Exclusion Criteria:

* children taking anti-parasitic drugs within the previous two weeks of stool sample collection .

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: samples will be collected from school children whose age is between 6-12 from different locations (cities and village).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of Feconomics technique which is a new ready to use kit for concentration of stool samples , for diagnosis of intestinal parasitic infections in children | 6 months following the startpoint of the study
  Comparing the sensitivity and specificity with traditional techniques i.e., direct smear and formalin ethyl acetate sedimentation technique for diagnosis of intestinal parasitic infections by examining stool samples from 100 patients, the number of cases with any intestinal parasite will be recorded.

IPD SHARING:
Plan to Share IPD: Undecided